CLINICAL TRIAL: NCT02768896
Title: Monitoring Brain Waves in Response to Visual and/or Auditory Stimulation in Parkinson's Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0182-16RMB
Record Dates: First submitted 2016-04-04; First posted 2016-05-11 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Baseline (No Intervention): Patients will walk naturally with EEG measuring brain waves
- Visual stimuli (Experimental): Patients will walk naturally with EEG measuring brain waves while seeing a grid through glasses
  Interventions: Behavioral: Baseline; Behavioral: visual stimuli
- Auditory stimuli (Experimental): Patients will walk naturally with EEG measuring brain waves while hearing an auditory stimuli
  Interventions: Behavioral: Baseline; Behavioral: Auditory stimuli
- Visual and auditory stimuli (Experimental): Patients will walk naturally with EEG measuring brain waves while seeing a grid through glasses and hearing an auditory stimuli simultaneously
  Interventions: Behavioral: Baseline; Behavioral: Visual and auditory stimuli

INTERVENTIONS:
Behavioral: Baseline — Patients will walk naturally with EEG measuring brain waves
  Arms: Auditory stimuli; Visual and auditory stimuli; Visual stimuli
Behavioral: visual stimuli — Patients will walk naturally with EEG measuring brain waves while seeing a grid through glasses
  Arms: Visual stimuli
Behavioral: Auditory stimuli — Patients will walk naturally with EEG measuring brain waves while hearing an auditory stimuli
  Arms: Auditory stimuli
Behavioral: Visual and auditory stimuli — Patients will walk naturally with EEG measuring brain waves while seeing a grid through glasses and hearing an auditory stimuli simultaneously
  Arms: Visual and auditory stimuli

SUMMARY:
Voltage fluctuation as a result of brain activity will be recorded into the computer using an EEG device.

DETAILED DESCRIPTION:
Patients with Parkinson's disease may have gait disturbances including freezing of gait. Visual and auditory stimuli may improve gait. Investigators will analyze brain wave during walking while giving the subject different stimuli.

The voltage fluctuation (in hundreds of microvolts) will be recorded using the EEG cap and amplifier into a computer.

ELIGIBILITY:
Inclusion Criteria:

• Patients with Parkinson's disease that are ambulatory and can sign a written informed consent

Exclusion Criteria:

* Patients with Parkinson's disease who are not ambulatory
* Patients with dementia
* Patients that are blind
* Patients that have severe hearing impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Voltage fluctuation resulting from brain activity after visual stimuli | One hour
  Change in brain wave activity after visual stimuli as compared with baseline measured in tens of micro-volts per second.
Voltage fluctuation resulting from brain activity after auditory stimuli | One hour
  Change in brain wave activity after auditory stimuli as compared with baseline measured in tens of micro-volts per second.
Voltage fluctuation resulting from brain activity after visual and auditory stimuli | One hour
  Change in brain wave activity after visual and auditory stimuli as compared with baseline measured in tens of micro-volts per second.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No